CLINICAL TRIAL: NCT06813547
Title: The Effect of Emotional Freedom Techniques and Virtual Reality Application Applied to Reduce the Fear of Childbirth on Attachment and Mental Well-being in Primiparous Pregnant Women
Brief Title: Emotional Freedom Techniques and Virtual Reality Application for Fear of Childbirth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sinem GUVEN Santur, Res. Assist., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Institute of Health Sciences
Record Dates: First submitted 2024-12-12; First posted 2025-02-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Fear of Childbirth; Mental Well-being; Attachment; Emotional Freedom Technique; Virtual Reality; Primiparous Pregnant Women
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional freedom techniques group (Experimental): Emotional Freedom Techniques (EFT) application group; Participants will receive EFT intervention once a week for four weeks, with pre- and post-assessment using scales and subjective experience units.
  Interventions: Behavioral: emotional freedom techniques
- Emotional freedom techniques + virtual reality group (Experimental): Emotional Freedom Techniques (EFT) and Virtual Reality (VR) application group; Participants will receive both EFT and VR interventions once a week for four weeks, with pre- and post-assessment using scales and subjective experience units.
  Interventions: Behavioral: emotional freedom techniques and virtual reality
- Control group (Other): Control group; Participants will receive standard antenatal care with pre- and post-assessment using scales and subjective experience units, but no EFT or VR intervention.
  Interventions: Behavioral: control group/ none intervention

INTERVENTIONS:
Behavioral: emotional freedom techniques — emotional freedom techniques
  Arms: Emotional freedom techniques group
Behavioral: emotional freedom techniques and virtual reality — emotional freedom techniques and virtual reality
  Arms: Emotional freedom techniques + virtual reality group
Behavioral: control group/ none intervention — None intervention
  Arms: Control group

SUMMARY:
Fear of labour in primiparous pregnant women is an important factor that directly affects the mother-infant relationship and the mental health of the mother. In this process, it is common for expectant mothers to experience feelings of uncertainty and anxiety about labour. Such intense fear of birth may weaken maternal attachment and make it difficult for her to establish a healthy emotional relationship with her baby. In addition, this fear may negatively affect the mother's mental well-being and increase the risk of depression and anxiety.

In this context, emotional liberation techniques (EFT) and virtual reality (VR) applications stand out as effective nonpharmacological methods used to reduce fear of childbirth in primiparous pregnant women. EFT is a technique that provides relaxation by touching the energy meridians that help the person to regulate negative emotions and cope with stress. SG, on the other hand, allows expectant mothers to interact with simulations similar to the real world in a virtual environment, providing therapeutic benefits through distraction, stress reduction and cognitive restructuring, allowing them to manage their fears about birth and enter the process more prepared. The use of SLT and SG, especially for primiparous pregnant women, can alleviate these women's anxiety about childbirth and enable them to approach the process in a safer and more conscious manner. Thus, it may also help to reduce the negative effects on the mother's postnatal attachment and mental health.

This study aims to examine the effects of SLT and SG practices on fear of childbirth, attachment and mental well-being, and to reveal the effects of these two methods on primiparous pregnant women. In this context, this study will fill the gap in the literature by providing a new perspective in clinical practice and antenatal education programmes and will make important contributions to increase antenatal attachment and mental well-being in primiparous pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* No verbal communication problems
* Primiparous pregnancy
* 32/0-38/0 weeks of gestation
* Having a single, viable foetus
* No psychiatric disorder
* No obstetric complications
* Absence of scar tissue or an obstacle to touch at the points of EFT application

Exclusion Criteria:

* Not wanting to continue the research
* Early labour

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Wijma Birth Anticipation/Fear Scale - Version A | 32-38 weeks of gestation
  The level of fear of labour will be assessed using a validated instrument, the Wijma Birth Anticipation/Fear Scale (Version A). Scores range from 0 to 165, with higher scores indicating higher levels of fear of labour.
Warwick-Edinburgh Mental Well-Being Scale - WEMWBS | 32-38 weeks of gestation
  Mental well-being will be measured using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS). Scores range from 14 to 70, with higher scores indicating higher mental well-being
Prenatal Mother-Infant Attachment Prenatal Mother-Infant Attachment Prenatal Mother-Infant Attachment | 32-38 weeks of gestation
  Maternal attachment to the unborn baby will be evaluated using the Prenatal Maternal Attachment Scale. Scores range from 21 to 84, with higher scores indicating stronger maternal attachment.
Subjective Unit Experience Scale | 32-38 weeks of gestation
  The scale, which was developed by Hartmann is utilised in EFT applications and enables the individual to categorise their own emotions by evaluating them with numbers. The SUE, a specific EFT instrument, is utilised to ascertain the intensity (degree) of the emotion experienced at the commencement and conclusion of the session. The scale is scored between -10 and +10, with negative numbers denoting negative/unpleasant experiences and positive numbers denoting positive/pleasant experiences.

SECONDARY OUTCOMES:
Demographic Characteristics of Participants | 32-38 weeks of gestation
  Age, education level, marital status, socioeconomic status, gestational week, and previous pregnancy history will be collected using a demographic information form.
  Group Comparability After Randomization Baseline demographic and clinical characteristics will be analyzed to ensure balance across groups after randomization.
  Subgroup Analysis Based on Age and Education Level Intervention effects will be examined across subgroups categorized by age and education level.
  Duration of Fear of Childbirth The duration of childbirth fear (in weeks or months) will be self-reported by participants.
  Previous Psychological Support History Participants' history of psychological support will be recorded via self-reported questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Özşahin, Dr, Study Director — Inonu University
Locations (1):
- Malatya Training and Research Hospital, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Even if the participants voluntarily agree to participate in the research in the country we live in, I cannot make this sharing because it is not legal to share the individual data of the participants.

REFERENCES:
- [Background] Hajesmaeel-Gohari S, Sarpourian F, Shafiei E. Virtual reality applications to assist pregnant women: a scoping review. BMC Pregnancy Childbirth. 2021 Mar 25;21(1):249. doi: 10.1186/s12884-021-03725-5. PMID 33765969
- [Background] Koo CH, Park JW, Ryu JH, Han SH. The Effect of Virtual Reality on Preoperative Anxiety: A Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Sep 29;9(10):3151. doi: 10.3390/jcm9103151. PMID 33003411
- [Background] Freitas JRS, Velosa VHS, Abreu LTN, Jardim RL, Santos JAV, Peres B, Campos PF. Virtual Reality Exposure Treatment in Phobias: a Systematic Review. Psychiatr Q. 2021 Dec;92(4):1685-1710. doi: 10.1007/s11126-021-09935-6. Epub 2021 Jun 26. PMID 34173160
- [Background] Guven Santur S, Ozsahin Z. The Effects of Emotional Freedom Techniques Implemented During Early Pregnancy on Nausea-Vomiting Severity and Anxiety: A Randomized Controlled Trial. J Integr Complement Med. 2024 Sep;30(9):858-868. doi: 10.1089/jicm.2023.0586. Epub 2024 Mar 27. PMID 38531058
- [Background] Maples-Keller JL, Yasinski C, Manjin N, Rothbaum BO. Virtual Reality-Enhanced Extinction of Phobias and Post-Traumatic Stress. Neurotherapeutics. 2017 Jul;14(3):554-563. doi: 10.1007/s13311-017-0534-y. PMID 28512692
- [Background] Bilgic G, Citak Bilgin N. Relationship Between Fear of Childbirth and Psychological and Spiritual Well-Being in Pregnant Women. J Relig Health. 2021 Feb;60(1):295-310. doi: 10.1007/s10943-020-01087-4. Epub 2020 Sep 19. PMID 32949330
- [Background] Aguilera-Martin A, Galvez-Lara M, Blanco-Ruiz M, Garcia-Torres F. Psychological, educational, and alternative interventions for reducing fear of childbirth in pregnant women: A systematic review. J Clin Psychol. 2021 Mar;77(3):525-555. doi: 10.1002/jclp.23071. Epub 2020 Oct 20. PMID 33078851
- [Background] Anderson CA, Gill M. Childbirth related fears and psychological birth trauma in younger and older age adolescents. Appl Nurs Res. 2014 Nov;27(4):242-8. doi: 10.1016/j.apnr.2014.02.008. Epub 2014 Feb 27. PMID 24726421
- [Background] Moller L, Josefsson A, Lilliecreutz C, Gunnervik C, Bladh M, Sydsjo G. Reproduction, fear of childbirth and obstetric outcomes in women treated for fear of childbirth in their first pregnancy: A historical cohort. Acta Obstet Gynecol Scand. 2019 Mar;98(3):374-381. doi: 10.1111/aogs.13503. Epub 2018 Dec 3. PMID 30431149
- [Background] Deliktas A, Kukulu K. Pregnant Women in Turkey Experience Severe Fear of Childbirth: A Systematic Review and Meta-Analysis. J Transcult Nurs. 2019 Sep;30(5):501-511. doi: 10.1177/1043659618823905. Epub 2019 Jan 17. PMID 30651038